CLINICAL TRIAL: NCT05075876
Title: An Open-Label, Randomized, Single-Center, Two-period, Two-sequence Cross-over Study to Assess the Bioequivalence of a Single 6-day Application of SP-01 (Granisetron Patch) Manufactured at Two Different Sites in Healthy Chinese Subjects
Brief Title: Bioequivalence Study in Healthy Chinese Subjects Comparing SP-01 (Granisetron Patch) Manufactured at Two Different Sites
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Solasia Pharma K.K. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SP-0105
Record Dates: First submitted 2021-09-21; First posted 2021-10-13 (Actual); Last update posted 2022-02-09 (Actual); Status verified 2022-02

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (SP-01-K) (Experimental): Application of SP-01 manufactured by Site K (SP-01-K) for 6 days followed by washout period for 21 days followed by application of SP-01 manufactured by Site A (SP-01-A) for 6 days
  Interventions: Drug: SP-01 manufactured by Site K (SP-01-K, Transdermal patch contained granisetron); Drug: SP-01 manufactured by Site A (SP-01-A, Transdermal patch contained granisetron)
- Group 2 (SP-01-A) (Active Comparator): Application of SP-01 manufactured by Site A (SP-01-A) for 6 days followed by washout period for 21 days followed by application of SP-01 manufactured by Site K (SP-01-K) for 6 days
  Interventions: Drug: SP-01 manufactured by Site K (SP-01-K, Transdermal patch contained granisetron); Drug: SP-01 manufactured by Site A (SP-01-A, Transdermal patch contained granisetron)

INTERVENTIONS:
Drug: SP-01 manufactured by Site K (SP-01-K, Transdermal patch contained granisetron) — Single application for 6 days
Drug: SP-01 manufactured by Site A (SP-01-A, Transdermal patch contained granisetron) — Single application for 6 days

SUMMARY:
This study is an open-label, single-center, two-period, two-sequence crossover study to assess the bioequivalence of SP-01 (Sancuso®: Granisetron Patch) manufactured at two different sites. Either the test product, namely SP-01-K, or reference product, namely SP-01-A, will be applied to the subject once in each period.

ELIGIBILITY:
Inclusion Criteria:

1. Han Chinese male or female subject, with all of his/her biological parents and grandparents are of Han Chinese ethnicity (who do not belong to any Chinese minorities)
2. Subject aged between 18 and 55 years, inclusive, at the time of signing the informed consent form
3. Body weight ≥ 45 kg and body mass index (BMI) of 18 to 25 kg/m2, inclusive.
4. Generally in good health with no clinically significant abnormality. Clinically insignificant abnormalities may be acceptable at the discretion of the investigator.
5. Female subject.

   * Non-childbearing potential
   * For female subject of childbearing potential who used (and/have their partner used) two acceptable contraceptive methods for at least 4 weeks prior to the first dose of study drug, and agree to use two contraceptive methods during the entire study period and within 3 weeks after the patch removal in Period 2. If abstinence is an alternative lifestyle, subject who is practicing abstinence and agree to practice abstinence throughout the above-mentioned periods may be included into the study.
6. Male subject.

   * If male subject has a female partner with childbearing potential, he has used (or has his partner used) two acceptable contraceptive methods for at least 4 weeks prior to the first dose of study drug, and must agree to use (or has his partner used) two contraceptive methods during the entire study period and within 3 weeks after the patch removal in Period 2. If abstinence is an alternative lifestyle, subject who is practicing abstinence and agree to practice abstinence throughout the above-mentioned periods may be included into the study.
7. Ability to understand the nature, scope and possible consequences of participation in the study
8. Willing to comply with the study procedures and restrictions
9. Willing to give written informed consent voluntarily

Exclusion Criteria:

1. Known significant allergic conditions to any medications in general, or to transdermal therapeutic systems (e.g. Elastoplast®) or medical adhesive tapes/dressings in particular.
2. Concurrent clinically significant conditions or known history of clinically significant conditions including but not limited to hepatobiliary & pancreatic, renal, urinary, respiratory, gastrointestinal, endocrine, cardiovascular, neurological, immunological, haematological, musculoskeletal, dermatological and/or psychiatric disorders.
3. Subject has estimated creatinine clearance ≤ 80 mL/min calculated by Cockcroft Gault formula prior to the first dose of study drug.
4. Subject has abnormal Alanine Aminotransferase (ALT) and/or Aspartate Aminotransferase (AST) values prior to the first dose of study drug and the abnormality, as determined by investigators, makes the subject not suitable for participation in the study.
5. Subject has history of uncontrollable migraine or headaches.
6. Subject has any skin conditions (e.g. tattoos, wounds, oily skin) or diseases (e.g. dermatological disorder) that may hinder clinical assessments on the upper lateral arm where the study drug is applied.
7. Any conditions or illnesses that in the opinion of the Investigator may jeopardize subjects or interfere with the interpretation of study results.
8. Has used any prescribed or over-the-counter medication, vitamins, herbal supplements, vaccines, and/or hormonal contraceptive pill/patch/injection within 14-day period (use of acetaminophen/paracetamol as sole active ingredient within 7 days) prior to the first dosing of the study drug (Day 1). Exceptions include topical medications or eye drops with no systemic action.
9. Participation in any clinical studies which involve the use of investigational medicinal product(s) within 3 months prior to the first dose of study drug.
10. Blood loss or donation of more than 450 ml within 3 months prior to the first dose of study drug.
11. Female subject who is lactating or has positive pregnancy test result prior to the first dose of study drug.
12. Has not constantly resided in Hong Kong or with recent significant change in lifestyle and habits, including diet and exercise.
13. Engaged in strenuous exercise within 14 days prior to the first dose of study drug or unwilling to stop strenuous exercise throughout the entire duration of the study.
14. Refuse to refrain from swimming, prolonged soaking in water (e.g. bathing), sauna or activities that cause excessive sweating when wearing a study patch.
15. Refuse to refrain from activities such as sunbathing or tanning using tanning bed/sunlamps that expose the application site to direct sunlight when wearing a patch and within 10 days after the patch removal.
16. Refuse to avoid scrubbing and shaving the patch application site from 48 hours prior to patch application and when wearing a patch.
17. Refuse to avoid application of creams, lotions or oils to the patch application site from 48 hours prior to patch application and when wearing a patch.
18. Refuse to abstain from consuming grapefruit or grapefruit-containing beverages from 48 hours prior to the first patch application until the last PK blood sampling on Day 11 in each period
19. Regular consumption of large quantities of xanthine-containing beverages such as coffee, tea, chocolate, cola or other caffeinated beverages, defined as more than 6 cups per day within 3 months prior to signing informed consent.
20. Refuse to restrict the consumption of xanthine-containing beverages to a maximum of 2 cups per day during screening and Day 12 to Day 25 of period 1, and refuse to abstain from consuming xanthine-containing beverages from 48 hours prior to patch application until the last PK blood sampling on Day 11 in each period.
21. Regular consumption of alcoholic beverages that exceeds 14 units per week (1 unit = 360 ml of beer; 150 ml of wine; 45 ml of distilled spirits) within 3 months prior to signing informed consent.
22. Refuse to restrict the consumption of alcoholic beverages to a maximum of 1 unit per day during screening and Day 12 to Day 25 of period 1, and refuse to abstain from alcoholic beverages from 48 hours prior to patch application until the last PK blood sampling on Day 11 in each period.
23. Regular tobacco smoking or using nicotine containing product of more than 3 cigarettes per day within 3 months prior to signing informed consent.
24. Refuse to abstain from tobacco smoking or using nicotine containing product from screening until Day 11 of Period 2.
25. History of substance (alcohol or illicit drugs) abuse/addiction in the past 5 years, or used illicit drugs 3 months prior to signing informed consent, or positive urine drug test and blood alcohol test prior to the first dose of study drug.
26. Subject has an immediate family member (e.g. spouse, parent/legal guardian, sibling or child) who is the study site or sponsor staff and directly involved with this study.
27. Any other concerns that the Investigator considers the subject not suitable for participation in the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2021-10-13 (Actual); Primary Completion 2021-12-03 (Actual); Study Completion 2021-12-03 (Actual)

PRIMARY OUTCOMES:
Maximum observed drug concentration (Cmax) | 11 days
  Maximum observed drug concentration in plasma
Area under the concentration-time curve (AUC) 0-t | 11 days
  Area under the plasma concentration-time curve from time zero to time t, where t is the last time point with non-zero concentration
AUC0-∞ | 11 days
  Area under the plasma concentration-time curve from time zero to time infinity

SECONDARY OUTCOMES:
Time to reach Cmax (Tmax) | 11 days
  Time to reach the maximum observed drug concentration in plasma
Terminal elimination rate constant (λZ) | 11 days
  Apparent terminal phase rate constant, where λZ is the magnitude of the slope of the linear regression of the log concentration versus time profile during the terminal phase
Elimination half-life (t1/2) | 11 days
  The time required for the observed drug concentration in plasma to reach half of its original value
Adverse event | 38 days
  Incidence of adverse events
Adhesion | 7 days
  Mean adhesion score, which is the average of adhesion scores of a subject in a period

CONTACTS AND LOCATIONS:
Overall Officials: Bernard Man Yung Cheung, Principal Investigator — Phase 1 Clinical Trials Centre, The University of Hong Kong
Locations (1):
- Phase 1 Clinical Trials Centre, The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No